CLINICAL TRIAL: NCT04717011
Title: Case Series Biomedical Study to Detect the Presence of SARS-CoV-2 in Semen of Patients Diagnosed With COVID-19 Disease
Brief Title: Case Series Study to Detect SARS-CoV-2 in Semen of COVID-19 Patients
Acronym: COVID-19CAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-COV-NA-20-05
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; COVID-19; Severe acute respiratory syndrome coronavirus 2; Semen
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR test — PCR test in two different semen samples from each patient: first with positive diagnosis for COVID-19 and the second after negative diagnosis for COVID-19.

SUMMARY:
A descriptive, clinical series, single-centre, national, biomedical study to determine the presence of SARS-CoV-2 in sperm samples from positive PCR patients for COVID-19 and to evaluate the presence of the virus in the sperm samples after a negative PCR for COVID-19

DETAILED DESCRIPTION:
In late December 2019, a new coronavirus strain emerged in China causing coronavirus disease 2019 (COVID19). Since then, COVID19 has become a global pandemic outbreak being declared a "public health emergency of international concern" by the International Health Regulations Emergency Committee of the WHO on January 30, 2020. The pandemic concerns to public worldwide but also to couples aiming to conceive through natural means or undergoing assisted reproductive technologies (ART). Different organizations including the American Society of Reproductive Medicine have recommended a precautionary approach. Therefore, new cycles for infertility patients as well as non-medically urgent gamete preservation treatments, such as social egg freezing, have been suspended in many countries. The decision to resume the In vitro fertilization (IVF) treatment make us to question if virus could be in gametes affecting couples and reproductive outcomes. The presence of the virus in sperm have contradictory results.

The present study aims to describe if there could be presence of virus in sperm samples of patients with positive diagnosis for COVID-19, and if so, if the virus turns negative on the sperm after the patient recovers and have a negative result for COVID-19. Also it aims to assess the presence of the virus in the seminal plasma and discern if it possible to disseminate it by sexual transmission.

An interim analysis is expected to be carried out once the 50% of the expected recruitment is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose written informed consent approved by the Ethics Committee (EC) has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
* Male age: 18 - 65 years, both included.
* COVID-19 positive result by PCR (including symptomatic and asymptomatic subjects).

Exclusion Criteria:

* Patients with severe symptoms or any other medical condition that is unstable or which, according to medical criteria, may put at risk the patient's safety and his compliance in the study
* Known medical history of azoospermia or anejaculation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include males diagnosed with COVID-19 by positive PCR with ages between 18-65. These patients will be recruited from all participant departments of the hospital and organized by the Quality and/or Occupational Safety department.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 semen result | 1 day
  PCR results in semen specimen samples with patient COVID-19 positive test

SECONDARY OUTCOMES:
SARS-CoV-2 semen result | 2-8 weeks
  PCR results in semen specimen samples with patient COVID-19 negative test

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simon, MD, PhD, Study Chair — Igenomix; Nasser Al-Asmar, PhD, Principal Investigator — Igenomix
Locations (1):
- Hospital Ruber Internacional, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No